CLINICAL TRIAL: NCT04822090
Title: Acute Human Parvovirus B19 Infection Triggers Immune-Mediated Transient Bone Marrow Failure Syndrome, Extreme Direct Hyperbilirubinemia and Acute Hepatitis in Patients With Hereditary Hemolytic Anemias: Multicenter Pathophysiological Study
Brief Title: Parvovirus B19 Infection in Hereditary Hemolytic Anemias Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ibrahim Yousef, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-21-02-23
Record Dates: First submitted 2021-03-22; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Parvovirus B19 Infection
Keywords: Parvovirus B19; Hereditary Hemolytic Anemias; Extreme Hyperbilirubinemia
MeSH Terms: conditions — Erythema Infectiosum; Anemia, Hemolytic, Congenital | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I: HHA patients with acute symptomatic HPV-B19 infection
  Interventions: Other: Supportive treatment with or without red cell transfusion/intravenous immune globulin (IVIG)
- Group II: HHA patients without acute symptomatic HPV-B19 infection

INTERVENTIONS:
Other: Supportive treatment with or without red cell transfusion/intravenous immune globulin (IVIG) — red cell transfusion; plasma exchange; renal replacement therapy; intravenous immunoglobulin. plasma exchange
  Groups: Group I

SUMMARY:
Although many studies investigated the prevalence and manifestations of HPV-B19 infection in patients with sickle cell anemia (SCA), thalassemia, and hereditary spherocytosis (HS) separately, there is limited information about the extent to which HPV-B19 infection leads to severe complications and chronic infection.

DETAILED DESCRIPTION:
HPV-B19 is the smallest single-stranded, linear DNA virus that causes human diseases. Exposure to respiratory secretions is the most common means of transmission of this virus. Infection is associated with a variety of manifestations ranging from asymptomatic to severe complications that depending on the host's hematological and immunological status. No prospective comparative studies investigated the risks associated with this pathogenic virus and predicted the disease course and morbidity among hereditary hemolytic anemia (HHA) patients classified by their underlying diseases.

Nobody has studied the underlying causes of the different and unusual presentations in acute symptomatic HPV-B19 infection in hereditary hemolytic anemias patients. So that, this first head-to-head study to compare thalassemia, sickle cell anemia (SCA), and spherocytosis (HS) patients presented with acute symptomatic HPV-B19 infection.

Studying the relationship between viremia, humoral immune response, and the underlying disease in patients presenting with acute symptomatic HPV-B19 infection should be useful for clarifying the undiagnosed pathophysiological mechanisms and other accessory factors to improve the diagnosis and management.

Moreover, early diagnosis of risk factors of unusual presentations of acute symptomatic HPV-B19 infection will be a useful tool for better treatment strategy, follow up and prognosis as well as prevent future complications

Patients admitted from haematology clinics and emergency departments of Sohag and Assiut University Hospitals for HHA-related complications or manifestations suggesting HHA were screened continuously between February 2018 to February 2020 for enrolment in this study and monthly followed for at least one-year and 3 years post HPV-B19 infection.

Design of the study

1. Patients

First 2 years, the candidate patients who will have evidence of HHA and/or will present with manifestations suggesting HHA and agree to comply with follow-up instructions will be screened for enrollment in this study and additional will be followed for at least one-year post-HPV-B19 infection. Patient data will be included demographics, relevant comorbidities, need for hospital admission, need for blood or plasma transfusion, renal replacement therapy or plasma exchange, hospital length of stay, completion of hospitalization (hospital discharge and death), cardiac events, neurological and respiratory events, type of treatments administered, and inflammatory laboratory parameters.

Diagnosis of HHA in the study patients

Laboratory investigations

1. Routine Biochemical Investigations Liver and renal function tests (LFTs), bilirubin, blood sugar, lipid, and indicated hormonal profiles will be performed on Cobas c 311& modular P auto analyzer (Roche Diagnostics, Mannheim, Germany), lactate dehydrogenase (LDH)

   : analysis will be done with Dimension Rx Max-Siemens & urine analysis, and albumin creatinine ratio will be performed for all patients.
2. Hematological analysis Complete blood count: peripheral blood samples will be withdrawn for diagnostic laboratory investigations and routine follow-up. 2- ml blood will be collected on potassium- ethylene diamine tetra-acetic acid (EDTA) anticoagulant coated tube for CBC using Cell-Dyn 3700, automated cell counter (Abbott diagnostic, Dallas, USA).

   Hereditary Hemolytic Anemia Diagnosis HHA will be suspected by clinical/family history of patient, examination, and laboratory tests including full complete blood count (CBC), calculation of red blood cells (RBCs) indices, corrected reticulocyte count, peripheral blood smear (PBS), iron study, total and direct bilirubin (TB, DB), increased serum LDH, decreased serum haptoglobin, and negative direct antiglobulin (Coomb's) test.

   Confirmation of HHA and identification of subtypes will be done by a series of specialized investigations as following:

   A. Diagnosis of hemoglobinopathy

   The protocol of Hb electrophoresis, sickle solubility testing, and studying Hb fractions with high-performance liquid chromatography (HPLC) will be used for the diagnosis of hemoglobinopathies, such as SCA and thalassemia as previously described.

   B. Diagnosis of RBC Membranopathy and Enzymopathy Hereditary red cell membrane disorders, such as HS and elliptocytosis will be identified by blood smear examination, red cell osmotic fragility test (OFT) with and without 24 hours incubation, acidified glycerol lysis test (AGLT), and RBC labeling with eosin-5'-maleimide (EMA) dye and subsequent measurement of RBC mean fluorescence intensity (MFI) by flowcytometry as previously described.

   Patients considered having HS will base on clinical and laboratory signs of chronic hemolysis, presence of spherocytes at PBS, plus two positive tests (OFT, AGLT, and EMA binding test) or at least one test with a family history of HS, and exclusion of other causes of secondary spherocytosis.

   All patients will be evaluated for RBC enzymes' activity, such as glucose-6-phosphate dehydrogenase (G6PD) to detect the coexistence of RBC enzymopathies and membranopathy.
3. Detection of HPV-B19 and HHA-Patients' Comparator Groups During the study period, any HHA-patient will have manifestations suggesting HPV-B19 infection (fever/ muscle pains /rash/ arthropathy/ lymphadenopathy/ rapid drop in Hb level and reticulocytopenia) and/or contact with a suspected case of erythema infectiosum will be investigated for anti-parvovirus B19 IgM and IgG immunoglobulin status. Those HPV-B19 seronegative will be retested 2 to 3 weeks later. HPV-B19 immunoglobulins (IgM and IgG) status will be determined by chemiluminescent immunoassays (CLIA) technology from (Diasorin, Saluggia, Italy). Additionally, serological tests for hepatitis, HIV, CMV, and EBV viruses will be done to exclude other recent viral infections. Blood cultures and sensitivity will be performed to exclude septicemia. The presence of signs, symptoms, HPV-B19 specific IgM, and absence of IgM of other viruses will be considered as proof of recent symptomatic HPV-B19 infection. Patients will be divided based on previous criteria into two groups.

Group I= HHA patients with acute symptomatic HPV-B19 infection, Group II= HHA patients without acute symptomatic HPV-B19 infection. Then group I patients will be subdivided according to underlying disease into three subgroups: Group Ia: HPV-B19(+)β-thalassemia, Group Ib: HPV-B19(+)HS, and Group Ic: HPV-B19(+)SCA.

The different presenting features of HPV-B19 infection, such as a number of cytopenias, acute kidney injury (AKI), hepatitis, and level of hyperbilirubinemia in group I will be compared. AKI will be diagnosed and classified according to the last guidelines. Extreme hyperbilirubinemia will be considered when total bilirubin >25 mg/dL. The clinical presentation at baseline was recorded.

7.4. Other Investigations The diagnosis of HPV-B19 extra-hematological manifestations, associated autoimmune disorders, cellular and humoral immune deficiencies will be determined using several methods such as detection of several autoantibodies, flowcytometry, serum immunoglobulins level.

Histopathological studies of BM, spleen, and liver biopsies will be done after patients' acceptance in restricted conditions and according to guidelines for an indication of biopsy as:

* BM aspiration and biopsy will be done for patients with persistent severe BMF non responded to treatment.
* Splenic biopsy from patients who will be submitted for elective splenectomy according to recommendations regarding splenectomy in HHA(13).
* Liver biopsy will be done for patients with persistently abnormal liver function with serological test positive to autoimmune or sclerosing cholangitis to differentiate the underlying disease for proper management.

Radiologic assessment by echocardiography, X-ray chest and long bones, and abdominal ultrasound will be routinely performed for screening all patients. The HHA patients with extreme hyperbilirubinemia or obstructive jaundice will be screened by magnetic resonance cholangiopancreatography (MRCP).

Group I patients will be monthly followed for at least one-year post HPV-B19 infection. Group II patients will be diligently followed for the time of writing this manuscript. During this period, complications, and laboratory profiles including BM aspiration if the patient had severe cytopenia, will be checked. All patients will be scanned by echocardiography and examined by ultrasound to view the gallbladder, kidneys, spleen, and liver size (cm). The events of interest will be recorded, such as bone marrow failure (BMF), spleen sequestration, chest pain, vaso-occlusive crisis, cholelithiasis, cholecystitis, and choledocholithiasis and transfusion frequency

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hereditary hemolytic anemias patients (age above 12 years) presented with signs and symptoms of hereditary hemolytic anemia (HHA) and admitted or treated in emergency departments or Hematology Units at Internal Medicine Departments of various university hospitals will be screened for enrollment in this study.

Exclusion Criteria:

* • Patients will be diagnosed with non-HHA as ( autoimmune hemolytic anemia, microangiopathic hemolytic anemia (MAHA), Wilson disease, paroxysmal nocturnal hemoglobinuria (PNH).

  * HHA-patients will refuse to consent to this study.
  * Serologic evidence of recent virus infection other than human parvovirus B19 (HPV-B19); hepatitis A (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), hepatitis E virus (HEV,) cytomegalovirus (CMV), Epstein-Barr virus (EBV), or positive test for HIV.
  * HHA patients with uncontrolled diabetes mellitus (DM).
  * HHA patients with a history of nephrotic syndrome or chronic kidney disease(CKD).
  * HHA patients with a history of treatment by immunosuppressive drugs.
  * HHA patients with clinical and laboratory evidence of relevant toxicity related to iron chelation.
  * HHA patients with severe systemic diseases (such as cardiovascular, renal, and hepatic disease) or surgical/medical conditions that might interfere with follow-up instructions.
  * HHA patients with a life expectancy of less than 1 year.
  * HHA patients with psychiatric disorders or a history of drug abuse,
  * Pregnant women will be also excluded.
  * Patients are not a candidate for investigation (Refusal

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HHA Patients will be classified according to of presence or absence of acute symptomatic HPV-B19 infection
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Number of hereditary hemolytic anemias (HHA) patients with symptomatic HPV-B19 infection | 2 years
  During the study period, any HHA-patient will have manifestations suggesting HPV-B19 infection (fever/ muscle pains /rash/ arthropathy/ lymphadenopathy/ rapid drop in (hemoglobin) Hb level and reticulocytopenia) and/or contact with a suspected case of erythema infectiosum will be investigated for anti-parvovirus B19 IgM and IgG immunoglobulin status. Those HPV-B19 seronegative will be retested 2 to 3 weeks later. HPV-B19 immunoglobulins (IgM and IgG) status will be determined by chemiluminiscent immunoassays (CLIA) technology from (Diasorin, Saluggia, Italy).
  The presence of signs, symptoms, HPV-B19 specific IgM, and absence of IgM of other viruses will be considered as a proof of recent symptomatic HPV-B19 infection. Patients will be divided based on previous criteria into two groups.
  Group I= HHA patients with acute symptomatic HPV-B19 infection, Group II= HHA patients without acute symptomatic HPV-B19 infection.
Common clinical manifestations of symptomatic HPV-B19 infection in patients with HHA | 2 years
  A questionnaire about the occurrence of. (Fever/ muscle pains /rash/ arthropathy / lymphadenopathy/ worsening of anemia/ Heart failure/ neuropathy) will be performed to determine the clinical manifestations of symptomatic HPV-B19 infection among patients with HHA.
Number of cytopenias | 2 years
  Complete blood count (CBC): peripheral blood samples will be withdrawn for diagnostic laboratory investigations and routine follow-up. 2- ml blood will be collected on potassium- ethylene diamine tetra-acetic acid (EDTA) anticoagulant coated tube for CBC using Cell-Dyn 3700, automated cell counter (Abbott diagnostic, Dallas, USA). The number of reticulocyte counts will be reported also.
Number of patients presenting with extreme hyperbilirubinemia during HPV-B19 infection | 2 years
  Measurement of direct and indirect bilirubin level which will be performed on Cobas c 311& modular P auto analyzer (Roche diagnostics, Mannheim, Germany).
  Extreme hyperbilirubinemia will be considered when total bilirubin >25 mg/dL.
Frequency of autoimmune bone marrow failure | 2 years
  The diagnosis of autoimmune bone marrow failure will be determined using several methods such as detection of
  1. Several autoantibodies (antinuclear antibodies (ANA), anti-double-stranded DNA (anti-dsDNA)), coombs test with pancytopenia and hypocellular bone marrow (BM)
  2. Detection of the percentage of lymphocytes subsets, cytotoxic T cells and T helper cells, and regulatory T cells in the bone marrow by flowcytometry
  3. Bone marrow aspiration if the patient had severe persistent cytopenia with histopathological studies of BM
Frequency of autoimmune hepatitis | Through study completion
  The diagnosis of autoimmune hepatitis (AIH) will be determined using AIH diagnosis last guidelines to diagnose and management of AIH in adults (.Revised Original Pretreatment Scoring System of the International Autoimmune Hepatitis Group) by:-
  1. Detection of autoimmune hepatitis antibodies and immunoglobulin G level
  2. Exclusion of other viral causes of hepatitis by serology and PCR of HAV, HBV, HCV, EBV, CMV
  3. Exclusion of Wilson disease by serum ceruloplasmin, 24-hour urinary copper,
  4. Exclusion of hemochromatosis by serum ferritin level
  5. Histopathological studies of liver biopsies will be done after patients' acceptance in restricted conditions and according to guidelines for indication of biopsy.
Frequency of renal involvement and acute kidney injury | Through study completion
  The diagnosis of acute kidney injury (AKI) using AKI diagnosis last guidelines (Kidney Disease: Improving Global Outcomes KDIGO) and renal involvement will be determined by:-
  1. Serum creatinine and blood urea
  2. Urine amount and analysis
  3. Albumin creatinine ratio
  4. Histopathological studies of renal will be performed according to indication.

SECONDARY OUTCOMES:
Number of patients with HPV-B19 reinfection during short term follow-up period (one year) | 1 year post HPV-B19 infection
  During the first year post-HPV-B19 infection, the number of patients with HPV-B19 reinfection will be reported.
  Group (I) patients with manifestations suggesting HPV-B19 reinfection will be investigated for anti-parvovirus B19 IgM and IgG immunoglobulin status and/or PCR. HPV-B19 immunoglobulins (IgM and IgG) status will be determined by chemiluminiscent immunoassays (CLIA) technology from (Diasorin, Saluggia, Italy) and will be compared to the level of IgM and IgG of the previous infection.
Frequency of HPV-B19 reinfection during 3 years follow-up period and COVID-19 outbreak | 3 years post HPV-B19 infection
  During the 3 years post HPV-B19 infection, the frequency of HPV-B19 reinfection among patients with HHA will be reported.
  HHA patients with manifestations suggesting HPV-B19 reinfection will be investigated for anti-parvovirus B19 IgM and IgG immunoglobulin status and/or PCR. HPV-B19 immunoglobulins (IgM and IgG) status will be determined by chemiluminiscent immunoassays (CLIA) technology from (Diasorin, Saluggia, Italy) and will be compared to the level of IgM and IgG of the previous infections.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Yousef, MD, PhD, Principal Investigator — , Faculty of Medicine, Sohag University
Locations (1):
- , Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No